CLINICAL TRIAL: NCT03636763
Title: Dipeptidyl Peptidase-IV Inhibitors, Risk Factor for Development of Bullous Pemphigoid? : Multicenter Retrospective Study in France and Switzerland
Brief Title: Dipeptidyl Peptidase-IV Inhibitors, Risk Factor for Development of Bullous Pemphigoid?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-29
Record Dates: First submitted 2018-08-16; First posted 2018-08-17 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Bullous Pemphigoid
MeSH Terms: conditions — Pemphigoid, Bullous | interventions — Research Design; Dipeptidyl-Peptidase IV Inhibitors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bullous pemphigoid and diabetes 2: patients with Bullous pemphigoid and diabete type 2 data report about gliptin exposure will be performed
  Interventions: Drug: data report
- diabete type 2: patients with diabetes type 2 data report about gliptin exposure will be performed
  Interventions: Drug: data report

INTERVENTIONS:
Drug: data report — the information "gliptin exposure" will be reported
  Other Names: gliptin

SUMMARY:
Bullous pemphigoid (BP) is the most common autoimmune bullous dermatosis. It mainly affects the elderly, and its cutaneous manifestations are extremely varied. Since the publication of the first case of PB associated with sulfasalazine in 1970, several drugs have been reported for their potential link with the development of PB. Recently, cases of PB associated with dipeptidyl peptidase-IV (DPP4) inhibitors, also known as gliptins, have been reported. DPP4 inhibitors are oral antidiabetic agents prescribed to patients with type 2 diabetes, as monotherapy, in combination with other oral antidiabetic agents or with insulin.

In recent years, an increasing number of cases have been published, describing the potential role of gliptins in PB induction. All these clinical cases and pharmacovigilance analyzes tend to show an increased risk of developing BP in case of gliptin exposure.

The main objective is to evaluate the risk of developing a PB under DPP4 inhibitor treatment, comparing cases of diabetic patients with BP, to matched diabetic controls for sex and age, from French departments. Endocrinology in a retrospective study from 1 January 2014 to 31 July 2016.

The study will be conducted using databases of clinical and histological records. The investigators will perform a retrospective 1: 2 case-control study comparing cases with type 2 diabetes and BP to matched diabetic controls for sex and age, randomly drawn from French endocrinology departments (Marseille La Conception ) and Switzerland (Bern), between January 1, 2014 and July 31, 2016. the investigators will compare gliptin exposure in the case-control group versus the control group, adjusting for potential confounding bias using models. logistic regression.

DETAILED DESCRIPTION:
Bullous pemphigoid (BP) is the most common autoimmune bullous dermatosis. It mainly affects the elderly, and its cutaneous manifestations are extremely varied. Since the publication of the first case of PB associated with sulfasalazine in 1970, several drugs (spironolactone, furosemide, chloroquine, beta-blockers and various antibiotics) have been reported for their potential link with the development of PB. Recently, cases of PB associated with dipeptidyl peptidase-IV (DPP4) inhibitors, also known as gliptins, have been reported. DPP4 inhibitors are oral antidiabetic agents prescribed to patients with type 2 diabetes, as monotherapy, in combination with other oral antidiabetic agents or with insulin.

Problem raised:

In recent years, an increasing number of cases have been published, describing the potential role of gliptins in PB induction. All these clinical cases and pharmacovigilance analyzes tend to show an increased risk of developing BP in case of gliptin exposure, but this hypothesis has not yet been confirmed by a quality controlled study.

Goal:

The main objective is to evaluate the risk of developing a PB under DPP4 inhibitor treatment, comparing cases of diabetic patients with BP, to matched diabetic controls for sex and age, from French departments. Endocrinology (Marseille La Conception) and Dermatologie (Marseille North, Marseille La Timone) and Swiss (Bern), in a retrospective study from 1 January 2014 to 31 July 2016.

Material and methods:

The study will be conducted in three university departments of Dermatology (Marseille North, Marseille La Timone, Bern), using databases of clinical and histological records. The investigators will perform a retrospective 1: 2 case-control study comparing cases with type 2 diabetes and BP to matched diabetic controls for sex and age, randomly drawn from French endocrinology departments (Marseille La Conception ) and Switzerland (Bern), between January 1, 2014 and July 31, 2016. The investigators will compare gliptin exposure in the case-control group versus the control group, adjusting for potential confounding bias using models. logistic regression.

Criteria for inclusion:

* Case: Patients from three university departments of Dermatology (Marseille North, Marseille La Timone, Bern) with type 2 diabetes, and a diagnosis of PB diagnosed for the first time between January 1, 2014 and July 31, 2016. The diagnosis of PB is based on compatible clinical presentation, compatible histology, positive direct immunofluorescence (IFD), and in some cases positive indirect immunofluorescence (IFI) and / or the presence of autoantibodies (BP180 and / or BP230) by ELISA.
* Witnesses: Patients from two university departments of Endocrinology (Marseille La Conception and Bern) with type 2 diabetes, and matched 1: 2 to cases for sex and age.

Exclusion criteria:

* Case: Patients with another bullous dermatosis, not meeting the inclusion criteria. Patients biopsied before consultation in University Hospital, or patients seen in private dermatology practices.
* Witnesses: Patients suffering at the time of inclusion of a chronic dermatosis, in particular of a bullous dermatosis.

ELIGIBILITY:
Inclusion Criteria:

Case: Patients from three university departments of Dermatology (Marseille North, Marseille La Timone, Bern) with type 2 diabetes, and a diagnosis of PB diagnosed for the first time between January 1, 2014 and July 31, 2016. The diagnosis of PB is based on compatible clinical presentation, compatible histology, positive direct immunofluorescence (IFD), and in some cases positive indirect immunofluorescence (IFI) and / or the presence of autoantibodies (BP180 and / or BP230) by ELISA.

- Witnesses: Patients from two university departments of Endocrinology (Marseille La Conception and Bern) with type 2 diabetes, and matched 1: 2 to cases for sex and age.

Exclusion Criteria:

Case: Patients with another bullous dermatosis, not meeting the inclusion criteria. Patients biopsied before consultation in University Hospital, or patients seen in private dermatology practices.

Witnesses: Patients suffering at the time of inclusion of a chronic dermatosis, in particular of a bullous dermatosis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from three university departments of Dermatology with type 2 diabetes and a diagnosis of PB diagnosed for the first time between January 1, 2014 and July 31, 2016
Sampling Method: Probability Sample
Enrollment: 183 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
numbers of patients exposed to gliptin | 3 years
  numbers of patients exposed to gliptin developing a Bullous pemphigoid

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — APHM
Locations (1):
- Assistance Publique Des Hopitaux de Marseille, Marseille, PACA, France